CLINICAL TRIAL: NCT05410353
Title: Managing Obesity by Leveraging Health Information Technology to Lower Cancer Risk
Brief Title: Choosing Healthy Activities and Lifestyle Management Through Portal Support
Acronym: CHAMPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20-07328-FB; 5R01CA267643-03 (NIH)
Record Dates: First submitted 2022-05-25; First posted 2022-06-08 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Weight Loss; Overweight and Obesity; Behavior, Health
Keywords: health information technology; electronic health record; patient portal
MeSH Terms: conditions — Weight Loss; Overweight; Obesity; Health Behavior

STUDY DESIGN:
Intervention Model Description: This is a 2-arm, parallel, randomized, controlled clinical trial. Eligible participants will be randomly assigned in a 1:1 ratio to either a behavioral weight loss intervention group delivered via Health IT with telephonic support (Active Intervention Group) or the Comparison Group. Because intervention delivery does not depend on clinic site, the study team has opted for a more powerful individual randomization over cluster randomization (but the team will potentially include clinic site as a grouping effect in the analysis).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomized portion of this protocol will employ a blinding design so that the CHAMPS study personnel and investigators who are collecting and assessing outcome data (i.e., weight) will not know a participant's group assignment status (blinded to assignment). Neither the participants, nor the study staff who provide the intervention, will be blinded to assignment. All participants will be asked not to reveal their CHAMPS study group assignment to blinded clinic personnel. All intervention-related information will be kept separately from outcome data and will not be accessible to blinded staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention Group (Experimental): Look AHEAD Intervention program adapted for delivery via Health IT modified for cultural and social norms applicable to different population groups
  Interventions: Behavioral: Active Intervention Group
- Comparison Group (Active Comparator): Look AHEAD DSE (Diabetes Support and Education) Comparison Group intervention adapted to be delivered via the EHR patient portal with telephonic support
  Interventions: Behavioral: Comparison Group

INTERVENTIONS:
Behavioral: Active Intervention Group — The 3 major intervention components are diet, physical activity, and the behavioral modification curriculum. Scheduled interactions are educational podcasts (a series of audiovisual, digital media files) paired with a follow-up phone counseling session with a trained behavioral interventionist. A patient portal message will be sent to participants when a new podcast is posted. Interactive sessions will be weekly (weeks 1-16), biweekly (weeks 17-24), and monthly (weeks 25-52). The goal for weight loss is ≥ 7% of initial weight over the course of 12 months. Participants will restrict caloric intake with the goal of 1,200-1,500 kcal/day for those weighing < 114 kg and 1,500-1,800 kcal/day for those weighing ≥ 114 kg. The physical activity goal will be for participants to gradually increase to 175-200 minutes of moderate-intensity activity per week by the 24th week. Participants will also be asked to self-monitor their dietary intake and physical activity using the "Lose It!" app.
  Other Names: Weight Loss; Adapted Look AHEAD ILI Group
  Arms: Active Intervention Group
Behavioral: Comparison Group — All participants in the Comparison Group will receive a mandatory 13 contacts per year including 3 informational sessions on nutrition, physical activity and social support and 10 contacts via patient portal or email regarding intervention topics. The Look AHEAD Comparison Group was designed to be realistic, achievable, and an acceptable intervention that encouraged optimal study retention.
  Other Names: Adapted Look AHEAD DSE Group
  Arms: Comparison Group

SUMMARY:
The study aims to randomize 250 participants to 1 of 2 arms: a.) an Active Intervention Group (based on the Look AHEAD* ILI) or b.) a Comparison Group (based on the Look AHEAD DSE Comparison group) to test the hypothesis that a multicomponent, multilevel behavioral weight loss intervention (Active Intervention Group) adapted for different population groups and delivered through Health Information Technology (Health IT) tools via the Electronic Health Record (EHR) patient portal, will result in significantly greater weight loss 12 months after enrollment compared to the Comparison Group.

*The Look AHEAD study was a multi-center, randomized clinical trial involving overweight and obese persons with type 2 diabetes, aimed to determine the effects on the cardiovascular outcomes of an intensive lifestyle intervention (ILI) for weight loss, in comparison to the diabetes support and education intervention (DSE).

DETAILED DESCRIPTION:
This project tests whether the adapted Look AHEAD Intensive Lifestyle Intervention (ILI) will result in significant weight loss when delivered through Health IT - EHR patient portal compared to a Comparison group (based on Look AHEAD DSE Comparison group). This project will be conducted in 2 stages: a formative assessment stage (Stage 1) and a clinical trial stage (Stage 2).

During Stage 1, we will modify the interactive technology-based Look AHEAD ILI that we already developed for the TARGIT study (Active Intervention group). We will also adapt the Look AHEAD Comparison condition (DSE group) for our Comparison condition. We will also optimize the protocol for acceptability in different populations and in a rural setting.

During Stage 2, we will randomly assign 250 participants to either the Comparison Group or the Active Intervention Group to address the primary aim of testing the hypothesis that a multicomponent, behavioral weight loss intervention delivered through Health IT - patient portal will lead to significantly greater weight loss 12 months after enrollment in the Active Intervention group compared with the Comparison group. Our Health IT-based intervention is potentially cost-effective and thus disseminable to any practice-based physician group with access to an EHR with a patient portal.

ELIGIBILITY:
Inclusion Criteria:

1. are ≥ 16 years old
2. are overweight or obese (BMI ≥ 25 kg/m2)
3. have access to the Internet via the computer or use a cellphone with a data-plan access
4. are patients at one of the participating practice sites
5. are willing to accept a random assignment, and
6. are from different population groups (racial / ethnic minority, lower socioeconomic status, or reside in a rural location).

Exclusion Criteria:

1. coronary or cerebrovascular disease events or vascular procedures within the past 6 months
2. certain medical conditions that put participants at high risk of adverse events or preclude exercising
3. uncontrolled psychiatric disorders
4. current substance abuse, including heavy alcohol use ≥ 5 drinks on the same occasion for ≥ 5 days in the past 30 days
5. a history of amputation or bariatric surgery or are planning to have bariatric surgery within the next 12 months
6. current weight loss medication use
7. malignancy within the last 5 years (except skin cancer)
8. plans to move out of the area during the next year
9. current participation in another clinical trial
10. pregnancy or breast feeding or are planning to become pregnant within the next 12 months, and
11. instances judged by the investigators' and primary care providers' discretion.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Relative percentage change in weight | 12 months
  This is calculated for each follow-up visit as ((weight at FU visit - baseline weight) / (baseline weight)) × 100%.

SECONDARY OUTCOMES:
Relationship of mutlitlevel determinants of health (screening tool) with weight change over time | 12 months
  How multilevel determinants of health, assessed via the Social Needs Screening Tool, relate to patient success with weight loss
Relationship of mutlilevel determinants of health (BRFSS) with weight change over time | 12 months
  How multilevel determinants of health, assessed via the Social Determinants of Health Questions Adapted from the Behavioral Risk Factor Surveillance System (BRFSS) 2017 Questionnaire, relate to patient success with weight loss
Relationship of multilevel determinants of health (z codes) with weight change over time | 12 months
  How multilevel determinants of health, assessed using z codes for Social Determinants of Health constructs abstracted from the Electronic Health Record using ICD -10 codes, relate to patient success with weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Karen Johnson, MD, Principal Investigator — University of Tennessee; Phyllis Richey, PhD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center / Department of Preventive Medicine, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will prepare and distribute a dataset maintaining confidentiality of individual participants. The final study analytical database will be processed according to HIPAA definitions for public data sharing and participant data will be de-identified using processes such as: removal of identifiers, translation of dates and ages to delta time values, and assignment of random study identifiers. A series of de-identified data files representing the final analytical data set will be available and provided in a standard format that is readable across a variety of applications and operating system platforms. Other documentation may include: data dictionary, data code book, valid variable ranges, protocol, MOP, intervention manual or programs, and any electronic versions of any paper forms that were used. The data release documentation will provide detailed, organized documentation of study variables and clear instructions on how to install and access the data.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Release and share the data no later than the acceptance of publication of the main finding of the final dataset
Access Criteria: Contact PI for access criteria